CLINICAL TRIAL: NCT03594409
Title: Frequency of Patho-morphological Classes of Gall Stones in Lahore, Pakistan
Status: Completed | Type: Observational
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principle investigator, Services Hospital, Lahore
Other Study IDs: s3
Record Dates: First submitted 2018-07-08; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Gallstone
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Biochemistry of gall stones — Analysis of gallstones is done to determine the biochemical types of gallstone like cholesterol stone, pigmented stones or mix stones

SUMMARY:
It is a cross sectional study in which we are tying to determine frequency of type of gall stones in our setup(Lahore, Pakistan).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with any sex age 1
2. 5 years and above
3. presenting to OPD with cholelithiasis -

Exclusion Criteria:

1. patients who develop gallstones after bariatric surgery
2. less than 15 years of age

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients selected from lahore and adjacent areas
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency of type of gallstones | 1 week
  primay outcome is to determine the frequency of biochemical classes of gallstones in lahore

CONTACTS AND LOCATIONS:
Overall Officials: Mahmmood Ayyaz, mbbs, fcps, Study Director — Services Hospital, Lahore
Locations (1):
- Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided